CLINICAL TRIAL: NCT00311194
Title: A Randomised, Controlled Trial of an Interactive CD-Program on 6 Months Readmission Rate in Patients With Heart Failure
Brief Title: Trial of an Interactive CD-Program on 6 Months Readmission Rate in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Heart Lung Foundation (Other)
Collaborators: The Council for Medical Health Care Research in South Sweden (Unknown); The Malmö University Hospital Research and Development Foundation (Unknown); The Skane County Councils Research and Development Foundation (Unknown); The NEPI Foundation (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: ABLM
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2006-04-05 (Estimated); Status verified 2002-05

CONDITIONS: Heart Failure
Keywords: Heart failure; Education; CD-ROM; Randomization; Hospitalization; Readmission; Death; Knowledge
MeSH Terms: conditions — Heart Failure; Death

INTERVENTIONS:
Behavioral: 6 months readmission rate to hospital

SUMMARY:
The purpose of this study is to determine whether extra education of patients with chronic heart failure can reduce 6 months readmission rate to hospital.

DETAILED DESCRIPTION:
The prevalence of heart failure (HF) has increased in the western world and is a major concern due to increasing prevalence and rising health care costs. The prognosis remains poor despite improvement in survival due to treatment with ACE-inhibitors and beta-receptor antagonists. HF has a high rate of readmission and hospitalisation. Some readmissions are ascribed to patients' lack of compliance, insufficient knowledge about diet, medication and symptoms of heart failure. Education of patients has become an important component in order to increase the patients' self-care and compliance. Intense education and counselling of patients is recommended in both European and American guidelines for HF.

Several systematic reviews of studies on strategies for improvement of outcomes of heart failure patients after discharge have been published, but very little emphasis has been put on methodological issues, e.g. methods of education. In most programs the methods and equipment used for education and information have only consisted of verbal and written material; computer-based tools seem to be relatively new.

Interactive CD-ROM programs for HF patients can increase patients' knowledge about heart failure and its treatment. However, no studies have examined the clinical outcome, e.g. rate of readmission.

Comparison: Extra educated patients (interactive CD-ROM education) compared to standard educated patients on readmission rate or death during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients treated for heart failure with left ventricular ejection fraction (LVEF) < 40 % at echocardiography or at least two of the criteria pulmonary rates, peripheral oedema, a third heart sound and signs of heart failure at chest X-ray.

Exclusion Criteria:

* Somatic disease or physical handicap with difficulties to communicate or handle the technical equipment, patients with only little knowledge in Swedish, patients with expected problems with compliance due to alcohol/drug abuse or major psychiatric illness, and participation in a trial.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 206
Dates: Start 1998-02; Study Completion 2002-07

PRIMARY OUTCOMES:
Readmission and death rate at 6 months' follow up.

SECONDARY OUTCOMES:
Knowledge regarding heart failure and its treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hans Liedholm, MD, PhD, Study Director — Drug and Therapeutics Committee; Agneta Björck Linné, B Pharm, PhD, Study Chair — Drug and Therapeutics Committee
Locations (1):
- Drug and Therapeutics Committee, Malmoe University Hospital, Malmo, Sweden

REFERENCES:
- [Background] Liedholm H, Linne AB, Agelii L. The development of an interactive education program for heart failure patients: the Kodak Photo CD Portfolio concept. Patient Educ Couns. 1996 Nov;29(2):199-206. doi: 10.1016/0738-3991(96)00902-0. PMID 9006236
- [Background] Linne AB, Liedholm H, Israelsson B. Effects of systematic education on heart failure patients' knowledge after 6 months. A randomised, controlled trial. Eur J Heart Fail. 1999 Aug;1(3):219-27. doi: 10.1016/s1388-9842(99)00041-0. PMID 10935668
- [Derived] Linne AB, Liedholm H. Effects of an interactive CD-program on 6 months readmission rate in patients with heart failure - a randomised, controlled trial [NCT00311194]. BMC Cardiovasc Disord. 2006 Jun 24;6:30. doi: 10.1186/1471-2261-6-30. PMID 16796760